CLINICAL TRIAL: NCT06628882
Title: Comparison of Infraclavicular Block and Wide-Awake Local Anesthesia With No Tourniquet for Hand Surgery: A Prospective Randomized Controlled Study
Brief Title: Comparison of Infraclavicular Block and Wide-Awake Local Anesthesia With No Tourniquet for Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selcan Akesen, Anesthesiology and Reanimation Specialist, Uludag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-19/21
Record Dates: First submitted 2024-06-24; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia, Local; Hand Deformity
Keywords: hand surgery; Anesthesia; WALANT
MeSH Terms: conditions — Hand Deformities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infraclavicular Block (Active Comparator): Patients were placed in the supine position with the head facing the opposite direction of the blocked side .After sterilizing the skin with povidone iodine, a linear ultrasound probe was sterilized and placed vertically over the infraclavicular fossa to visualize the axillary artery and the lateral, medial, and posterior cords of the brachial plexus. Using an 80 mm long 21G Stimuplex1 needle, a mixture of 10 cc 0.5% bupivacaine (BUPIVON® liquid 5%, On Pharma, Istanbul, Turkey)and 2% lidocaine(JETOKAIN® liquid Adeka Pharma, Istanbul, Turkey) was injected around the three cords with intermittent aspiration for control purposes.
  Interventions: Procedure: Infraclavicular Block
- Wide-Awake Local Anesthesia with No Tourniquet (Experimental): The WALANT solution was prepared as follows: 50 mL of 1 mg/1 mL epinephrine + 2% lidocaine(JETOKAIN® liquid Adeka Pharma, Istanbul, Turkey) + 39 cc of 0.9% isotonic NaCl + 10 mL of 8.4% sodium bicarbonate . The surgical area was sterilized with polyvinyl iodine. Using a 27-gauge syringe, the solution was applied around the incision site, either from a single point or several different points, until whitening of the skin was observed. Care was taken not to exceed the maximum dose of 7 mg/kg. The surgical procedure began 20-30 minutes after the application of the WALANT technique.
  Interventions: Procedure: Wide-Awake Local Anesthesia with No Tourniquet

INTERVENTIONS:
Procedure: Infraclavicular Block — types of anesthesia used in upper extremity surgeries
  Arms: Infraclavicular Block
Procedure: Wide-Awake Local Anesthesia with No Tourniquet — types of anesthesia used in upper extremity surgeries
  Arms: Wide-Awake Local Anesthesia with No Tourniquet

SUMMARY:
The patients were randomized into the WALANT and ICB groups. The pain levels of the patients before, during, and after surgery were queried and recorded using the visual analog scale (VAS). Their satisfaction levels were evaluated using a Likert scale. The duration of anesthesia administration, onset of the anesthesia effect, additional intraoperative analgesic needs, total duration of the anesthesia effect, postoperative analgesic needs, length of hospital stay, total surgical duration, hospitalization costs, and complications were evaluated.

DETAILED DESCRIPTION:
The inclusion criteria were patients between the ages of 18 and 70, an American Society of Anesthesiologists (ASA) physical status classification of I, II, or III, surgery planned for a single indication, and a surgery duration of between 20 and 60 minutes. The exclusion criteria were patients with an ASA classification >III, patients with planned bilateral surgery, patients with a local infection, patients with a neurological disorder affecting the same upper extremity, patients with a history of allergy to local anesthetic drugs, patients with a history of opioid use in the previous month, and patients who were unable to understand the study and answer the questions adequately.

WALANT: The WALANT solution was prepared as follows: 50 mL of 1 mg/1 mL epinephrine + 2% lidocaine + 39 cc of 0.9% isotonic NaCl + 10 mL of 8.4% sodium bicarbonate [11]. The surgical area was sterilized with polyvinyl iodine. Using a 27-gauge syringe, the solution was applied around the incision site, either from a single point or several different points, until whitening of the skin was observed. Care was taken not to exceed the maximum dose of 7 mg/kg. The surgical procedure began 20-30 minutes after the application of the WALANT technique. Figure 1 shows patients for whom the WALANT technique was administered..

ICB: Patients were placed in the supine position with the head facing the opposite direction of the blocked side .After sterilizing the skin with povidone iodine, a linear ultrasound probe was sterilized and placed vertically over the infraclavicular fossa to visualize the axillary artery and the lateral, medial, and posterior cords of the brachial plexus. Using an 80 mm long 21G Stimuplex1 needle, a mixture of 10 cc 0.5% bupivacaine and 2% lidocaine was injected around the three cords with intermittent aspiration for control purposes. Figure 2 shows patients who underwent the ICB procedure.

Clinical evaluation: Patients who could not achieve sufficient pain control were either sedated or switched to general anesthesia and were excluded from the study. The pain levels of the patients before, during, and after surgery were queried and recorded using the visual analog scale (VAS). The patients were asked whether they would prefer the same anesthesia method if another surgery were planned, and their satisfaction levels were evaluated using a Likert scale, where 1 indicated low levels of satisfaction, and 4 denoted high levels of satisfaction. The duration of anesthesia administration, onset of the anesthesia effect, intraoperative additional analgesic needs, total duration of the anesthesia effect, postoperative analgesic needs, length of hospital stay, total surgical duration, and complications were evaluated. The hospitalization costs (including the cost of drugs and anesthesia materials) of the WALANT and ICB groups were calculated and compared.

ELIGIBILITY:
Inclusion Criterias:

* American Society of Anesthesiologists (ASA) physical status classification of I, II, or III,
* surgery planned for a single indication
* surgery duration of between 20 and 60 minutes.

Exclusion Criterias:

* patients with an ASA classification >III,
* patients with planned bilateral surgery,
* patients with a local infection,
* patients with a neurological disorder affecting the same upper extremity,
* patients with a history of allergy to local anesthetic drugs,
* patients with a history of opioid use in the previous month,
* patients who were unable to understand the study and answer the questions adequately

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
the visual analog scale (VAS) | before surgery
  pain score - (0-10 point - higher scores mean worse)
the visual analog scale (VAS) | during surgery
  pain score - (0-10 point - higher scores mean worse)
the visual analog scale (VAS) | after surgery (Day 1)
  pain score - (0-10 point - higher scores mean worse)

SECONDARY OUTCOMES:
Likert scale(0-5 points) | after surgery (Day 0)
  levels of satisfaction (0-5 point - higher scores mean better)
Likert scale(0-5 points) | after surgery (Day 1)
  levels of satisfaction (0-5 point - higher scores mean better)

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No